CLINICAL TRIAL: NCT04387045
Title: Association of Perceived Stress and Negative Thoughts With Metabolic Biomarkers and Inflammatory Diseases in People With Type 2 Diabetes Mellitus and Healthy Subjects
Brief Title: Perceived Stress and Negative Thoughts With Biomarkers in People With Type 2 Diabetes Mellitus and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Carlos López Marquez (Other)
Responsible Party: Sponsor-Investigator, Francisco Carlos López Marquez, Director of Biomedical research center, Faculty of Medicine, Torreón unit., Universidad Autonoma de Coahuila
Organization: Universidad Autonoma de Coahuila (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C.B/02-01-17
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Depression; Stress; Negative thoughts
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guilty feelings (Experimental): Write for 20 minutes about a situation that in the participant's past life has caused feelings of guilt.
  Interventions: Behavioral: Guilty feelings
- Neutral feelings (Placebo Comparator): Write for 20 minutes about a situation that in the participant's past life has caused neutral feelings.
  Interventions: Behavioral: Guilty feelings

INTERVENTIONS:
Behavioral: Guilty feelings — Participants write for 20 minutes about situations that have caused them feelings of guilt throughout their lives.

SUMMARY:
The purpose of this study is to determine the effect of measured and induced negative feelings on glucose, tumor necrosis factor alpha, and cortisol levels in healthy participants and participants with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Depression and Diabetes are two pathologies that are frequently comorbid. Stress and negative thoughts are part of both. The biological correlates of psychological and emotional life are not yet fully clarified, so in this study we wonder about the association between tumor necrosis factor alpha, cortisol, and peripheral glucose levels with depression stress, measured negative thoughts, and induced guilt.This is a randomized intervention study. At baseline, participants complete the Beck Depression Inventory, the Automatic Negative Thoughts Scale (ATQ-N), and the Perceived Stress Scale (PSS-14). The intervention consists of a written task about situations that involved feelings of guilt or neutral situations. Saliva and dextrostix samples are taken before the 20-minute written task, at the end, dextrostix and saliva samples are performed again, finally a blood sample is taken.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent.
* 30 to 65 years of age.
* Current diagnosis of Diabetes mellitus type 2 without diabetic foot.
* Healthy volunteers.
* Ability to read and write.

Exclusion Criteria:

* Other current or past chronic disease diagnoses.
* Current use of antidepressants or other psychiatric medications.
* Steroid medication.
* Consumption of tobacco or alcohol in the last 24 hours.
* Previous diagnosis of autoimmune diseases

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Glucose levels | Sample collection is two times during a single day for each participant, with an interval of 20 minutes. Since it will be measured in fasting, it will take place between 8:00 a.m. and 9:00 a.m.
  mg/dL
Salivary cortisol | Sample collection is two times during a single day for each participant, with an interval of 20 minutes. Since it will be measured in fasting, it will take place between 8:00 a.m. and 9:00 a.m.
  mg/dL
Salivary Tumor Necrosis Factor alpha | Sample collection is two times during a single day for each participant, with an interval of 20 minutes. It will take place between 8:00 a.m. and 9:00 a.m.
  mg/dL

SECONDARY OUTCOMES:
Perceived stress | This variable is measured in a single day and represents the week prior to the study.
  Perceived stress scale (PSS-14), range 0-40.Higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Negative thoughts | This variable is measured in a single day and represents the month prior to the study.
  Automatic negative thoughts scale (ATQ-N), range 0-90. Higher scores mean a worse outcome (more negative thoughts).
Depression | This variable is measured in a single day and represents the week prior to the study.
  Beck's Depression Inventory, range 0-63. Higher number indicating more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco C. López Marquez, PhD, Principal Investigator — Universidad Autonoma de Coahuila, Centro de investigación Biomédica
Locations (1):
- Facultad de medicina De la UADEC Unidad Torreón, Torreón, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: No